CLINICAL TRIAL: NCT05911607
Title: Influence of Photobiomodulation Therapy (PBMT) as an Adjunctive Therapy in Alveolar Socket Preservation Preceding Dental Implant Placement
Brief Title: PBMT Influence on Alveolar Socket Preservation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamad Anwar Abd-Elhaleem Othman, Principal investigator, PhD candidate, researcher in National Institute of Laser Enhanced Sciences., Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2905561312919
Record Dates: First submitted 2023-06-02; First posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Extraction Socket Healing
MeSH Terms: interventions — Low-Level Light Therapy

STUDY DESIGN:
Intervention Model Description: Comparing between 2 laser' effect on extraction socket healing
Who Masked: Participant
Masking Description: Histological examination
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Red Laser (Active Comparator): Photobiomodulation using nm Diode.
  Interventions: Procedure: Low power laser
- Infrared Laser (Active Comparator): Photobiomodulation using nm Diode.
  Interventions: Procedure: Low power laser

INTERVENTIONS:
Procedure: Low power laser — Phototherapy for extraction sockets using two different lasers.

SUMMARY:
Goal of this study is to compare between the effect of two different low power lasers on extraction socket healing.

DETAILED DESCRIPTION:
After molar tooth extraction, 6 Low power (PBMT) laser sessions.

Evaluation:

Visual Radiographic Histological

ELIGIBILITY:
Inclusion Criteria:

* Fit for implant rehabilitation.
* Acceptable oral hygiene.
* Willingness to attend 6 visits within 15 days of extraction.

Exclusion Criteria:

* Uncontrolled diabetes.
* Sub optimal oral hygiene.
* Heavy smoker.

Ages: 30 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-09-15 (Actual)

PRIMARY OUTCOMES:
Radiographic socket dimensions | 3 months
  Alveolar Socket surface area measured on Cone Beam Computerised Tomography

SECONDARY OUTCOMES:
Soft tissue healing | 15 days
  Landry, Turnbull, Howley healing index; scoring from 1 to 5 where 1 represents very poor healing while 5 denotes perfect healing.
Histological examination | 3 months
  Histological examination of bone samples

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Ab Zaky, Study Director — National Institute of Laser Enhanced Sciences, Cairo University
Locations (1):
- National Institut of laser enhanced sciences, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rosero KAV, Sampaio RMF, Deboni MCZ, Correa L, Marques MM, Ferraz EP, da Graca Naclerio-Homem M. Photobiomodulation as an adjunctive therapy for alveolar socket preservation: a preliminary study in humans. Lasers Med Sci. 2020 Oct;35(8):1711-1720. doi: 10.1007/s10103-020-02962-y. Epub 2020 Jan 22. PMID 31970564